CLINICAL TRIAL: NCT06328140
Title: Sleep Quality, Cognitive Performance, and Computerized Cognitive Training Comparison of Patients Treated With Lurasidone vs.Patients With Major Depression Receiving Selective Serotonin Reuptake Inhibitor(SSRI) Treatment as Usual
Brief Title: Sleep Quality, Cognitive Performance, and Computerized Cognitive Training
Status: Withdrawn | Type: Observational
Why Stopped: we were unable to recruit participants according to the original protocol specifications. The sponsor would not allow for a modification so the study was stopped.
Sponsor: George West Mental Health Foundation d/b/a Skyland Trail (Other)
Collaborators: Sumitomo Pharmaceuticals America (Industry)
Responsible Party: Sponsor
Other Study IDs: Skyland 001
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-03

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Psychosis
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lurasidone Treatment: Patients with bipolar disorder or psychotic disorders for whom lurasidone is a US Food and Drug Administration (FDA)-approved treatment.
  Patients will be treated with a daily dose of 40-80 mg./day for schizophrenia and 30-60 mg./day for bipolar disorder.
  Interventions: Drug: Lurasidone
- Treatment as usual for major depression: Patients with major depression will received treatment with antidepressant treatments that are approved by the US FDA for treatment of major depression. All dosing will be required to be consistent with the FDA approved package insert.
  Interventions: Drug: FDA Approved antidepressant treatment

INTERVENTIONS:
Drug: Lurasidone — Daily medication treatment
  Groups: Lurasidone Treatment
Drug: FDA Approved antidepressant treatment — Daily treatment with an FDA approved antidepressant
  Other Names: Any FDA Approved antidepressant
  Groups: Treatment as usual for major depression

SUMMARY:
Poor sleep quality is common in neuropsychiatric conditions and some of the problems associated with poor sleep at night may be due to medication side effects or reduced efficacy of certain treatments. Poor sleep quality has been implicated in cognitive impairments, with the sleep quality to cognition association so strong that specialized assessments have been developed to examine the subjective association between poor nighttime sleep and daytime cognitive impairment.

Computerized cognitive training (CCT) is a training procedure designed to build cognitive skills, with a goal of improvement of functional outcomes. CCT is also a learning-based approach and previous studies have shown that successful CCT interventions lead to changes in brain circuitry. It is also known, however, that many cases who are treated with CCT fail to make treatment-related gains. Recent studies have suggested that this may be associated with failures to engage in the training procedures, which could be related to sleep related impairments.

Increased anticholinergic load can also substantially disrupt the process of training related gains directly. Antihistaminergic effects, common to many antidepressant and antipsychotic medications, can lead to daytime sedation and sleepiness, which both interferes with treatment but also interferes with nighttime sleep as well

In previous clinical trials, Lurasidone was associated with reductions in sleepiness and with cognitive gains that exceeded practice effects. One viable hypothesis is that Lurasidone has both direct beneficial effects on cognition and substantial indirect benefits, due to the lack of histamine receptor occupancy, lack of anticholinergic effects, and direct promotion of positive nighttime sleep outcomes.

Thus, a broad-spectrum naturalistic comparison of Lurasidone-treated patients with patients treated with other medications is proposed. This would include examining the level of engagement in CCT treatment, measurement of CCT training gains, and relating engagement and training gains with concurrent sleep quality, measured by actigraphy.

DETAILED DESCRIPTION:
Poor sleep quality is common in neuropsychiatric conditions and some of the problems associated with poor sleep at night may be due to medication side effects or reduced efficacy of certain treatments.

These impairments in daytime cognition seem most significant in areas relevant to daytime learning and nighttime memory consolidation, which has important implications for the success of rehabilitation focused psychiatric treatments. These treatments are learning based and functional and social skills are trained with teaching, which cannot be successful in the presence of significant memory consolidation problems. Reduced levels of slow wave sleep are likely to lead to problems in the consolidation of information presented for learning.

Computerized cognitive training (CCT) is a training procedure designed to build cognitive skills, with a goal of improvement of functional outcomes. CCT is also a learning-based approach and previous studies have shown that successful CCT interventions lead to changes in brain circuitry. It is also known, however, that many cases who are treated with CCT fail to make treatment-related gains. Recent studies have suggested that this may be associated with failures to engage in the training procedures, which could be related to sleep related impairments. These impairments could lead either to failures to concentrate during the daytime or failures to consolidate at night. As a result, the commonly expected benefits on neuroplasticity associated with CCT may be interrupted by poor sleep and this may lead to reduced benefits associated with combined skills training and CCT interventions.

In addition to the adverse effects of impaired sleep on consolidation and daytime alertness, there are multiple ways that these processes can be disrupted pharmacologically through several different factors. Increased anticholinergic load can substantially disrupt the process of training related gains directly. Antihistaminergic effects, common to many antidepressant and antipsychotic medications, can lead to daytime sedation and sleepiness, which both interferes with treatment but also interferes with nighttime sleep as well.

In a previous study, treatment with Quetiapine was previously found to induce substantial sleepiness and was associated with essentially no practice related improvements in cognition across 4 assessment time periods In contrast, Lurasidone was associated with reductions in sleepiness and with cognitive gains that exceeded practice effects. Thus, some of the differences in cognitive performance between quetiapine and Lurasidone could be due to sleep disturbance, in addition to the intrinsic benefits of lurasidone on cognition. One viable hypothesis is that Lurasidone has both direct beneficial effects on cognition and indirect benefits, due to the lack of histamine receptor occupancy, lack of anticholinergic effects, and direct promotion of positive nighttime sleep outcomes.

Thus, a broad-spectrum naturalistic comparison of Lurasidone-treated patients with patients treated with other medications is proposed. This would include baseline cognitive performance, measurement of treatment-related gains, and wearable devices.

The assessments goals would be to measure nighttime sleep, engagement in CCT, and cognitive gains over the study period. The primary outcome is cognitive gains with training over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic Criteria
* Patients with major depression or bipolar disorder will have baseline Brief Assessment of *Cognition (BACS) composite scores of 0.5 Standard deviations (SD) below normative (0.0) standards
* Patients with schizophrenia spectrum conditions will have baseline BACS composite scores 1.0 SD below normative (0.0) standards
* Able and willing to give informed consent
* Expected length of stay at least 8 weeks.

Exclusion Criteria:

* Symptoms Attributed to neurological Causes, including stroke or seizure disorder
* Sensory impairments precluding CCT
* Current treatment with vortioxetine or tricyclic antidepressants
* Patients with mood disorders will be excluded if they have BACS composite scores more than 2.5 SD below normative (0.0)standards Patients with schizophrenia spectrum conditions will be excluded if they have BACS composite scores more than 3.0 SD below normative (0.0) standards

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sampled from consecutive admissions to residential treatment at Skyland Trail.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Improvement in Cognitive Performance | Baseline to 8 weeks of treatment
  Composite Score on the Brief Assessment of Cognition: Standard score with population mean of 0 and Standard deviation of 1.0. Range is from -4.0 to 4.0; higher scores reflect better performance

SECONDARY OUTCOMES:
Training Engagement in Cognitive training | Baseline to 8 weeks of treatment
  Numbers of levels mastered per training day
Nighttime sleep measured with actigraphy | Baseline to 8 weeks of treatment
  Minutes of daily sleep indexed by a Fit-Bit Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Ben W Hunter, MD, Principal Investigator — Skyland Trail
Locations (1):
- George West Mental Health Foundation, DBA Skyland Trail, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harvey PD, Siu CO, Loebel AD. Change in daytime sleepiness and cognitive function in a 6-month, double-blind study of lurasidone and quetiapine XR in patients with schizophrenia. Schizophr Res Cogn. 2016 Jun 2;5:7-12. doi: 10.1016/j.scog.2016.05.002. eCollection 2016 Sep. PMID 28740811
- [Background] Harvey PD, Balzer AM, Kotwicki RJ. Training engagement, baseline cognitive functioning, and cognitive gains with computerized cognitive training: A cross-diagnostic study. Schizophr Res Cogn. 2019 May 13;19:100150. doi: 10.1016/j.scog.2019.100150. eCollection 2020 Mar. PMID 31832340